CLINICAL TRIAL: NCT00033475
Title: Cytotoxic T Cell Therapy for Post Transplant Lymphoproliferative Disease: Randomized Controlled Trial in Transplant Recipients
Brief Title: Reduced Immunosuppressive Therapy With or Without Donor White Blood Cells in Treating Patients With Lymphoproliferative Disease After Organ Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069288; CRUK-EBV-CTL; LCMV-CTL; EU-20057
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2025-09

CONDITIONS: Lymphoproliferative Disorder
Keywords: post-transplant lymphoproliferative disorder
MeSH Terms: conditions — Lymphoproliferative Disorders

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes

SUMMARY:
RATIONALE: Some types of lymphoproliferative disease are associated with Epstein-Barr virus. Combining reduced immunosuppressive therapy with donor white blood cells that have been treated in the laboratory to kill cells infected with Epstein-Barr virus may be an effective treatment for lymphoproliferative disease.

PURPOSE: Randomized phase III trial to compare the effectiveness of reducing immunosuppressive therapy with or without donor white blood cells in treating patients who have Epstein-Barr virus-associated lymphoproliferative disease after organ transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of treatment with partially HLA-matched allogeneic cytotoxic T cells and reduction of immunosuppression, in terms of survival rate and time to remission in patients with Epstein-Barr virus-associated B-cell lymphoproliferative disease after solid organ transplantation.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to transplanted organ type and transplant center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo sliding-scale reduction of immunosuppressive drugs from 1 of 5 regimens at physician's discretion. Patients then receive partially HLA-matched allogeneic cytotoxic T cells IV over 5 minutes once weekly for a total of 4 weeks.
* Arm II: Patients undergo reduction of immunosuppression as in arm I alone. Patients are followed monthly for 6 months and then every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of post-transplant lymphoproliferative disease (PTLD) after solid organ (heart, heart/lung, liver, liver/gut, pancreas, or kidney) transplantation

  * Epstein-Barr virus-positive tumor
  * Newly diagnosed disease
* Measurable disease by clinical methods or radiography
* Must have partially matched donor cytotoxic T cells (CTL) available
* No known panel reactivity to any of the HLA types of CTL available for therapy

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Karnofsky 20-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior therapy for PTLD
* No concurrent antiviral drugs (e.g., acyclovir or ganciclovir) for PTLD

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2001-03-01 (Actual)

PRIMARY OUTCOMES:
Complete response
Partial response
Stable disease
Progressive disease
Time to complete remission
Survival at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy H. Crawford, MD, Study Chair — University of Edinburgh
Locations (12):
- United Kingdom (12):
  - Birmingham Children's Hospital, Birmingham, England
  - Papworth Hospital, Cambridge, England
  - Royal Free and University College Medical School, London, England
  - King's College Hospital, London, England
  - Wythenshawe Hospital, Manchester, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Northern General Hospital, Sheffield, England
  - Institute of Cancer Research - UK, Sutton, England
  - Royal Infirmary of Edinburgh at Little France, Edinburgh, Scotland
  - University of Edinburgh, Edinburgh, Scotland
  - University of Edinburgh Laboratory for Clinical and Molecular Virology, Edinburgh, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland